CLINICAL TRIAL: NCT06948461
Title: An Adaptive Basket Trial to Evaluate Efficacy of Lyophilized Fecal Microbiota Therapy in Management of Irritable Bowel Syndrome-diarrhea Predominant or Prevention of Recurrent Clostridioides Difficile Infection
Brief Title: A Flexible Clinical Trial to Test if Freeze-dried Fecal Microbiota Therapy Helps Treat Diarrhea-predominant Irritable Bowel Syndrome or Prevent Recurring C. Difficile Infections.
Acronym: ORAL-LYO-FMT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaPlanter Technologies Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Basket ORAL-LYO-FMT Trial
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Irritable Bowel Syndrome, Diarrhea-Predominant (IBS-D); Recurrent Clostridioides Difficile Infection (rCDI); Fecal Microbiota Therapy (FMT); Irritable Bowel Syndrome (IBS); Clostridioides Difficile Infection
Keywords: IBS; Irritable bowel syndrome; rCDI; Fecal Microbiota Therapy; FMT; Gut Health; CDI; Clostridioides difficile infection, Recurrent
MeSH Terms: conditions — Irritable Bowel Syndrome; Clostridium Infections; Recurrence

STUDY DESIGN:
Intervention Model Description: This trial will use both a basket trial design and a parallel Simon two-stage design to reduce the time and costs to determine whether ORAL-LYO-FMT is effective and safe for IBS-D, and in prevention of additional recurrence of CDI for primary or rCDI.
  Basket trials are an innovative trial design that has been developed as an efficient way to determine safety and efficacy of experimental therapeutics across multiple patient populations and diseases. Basket trials assess the effectiveness of a drug based on its mechanism of action rather than the underlying disease. This type of trial design is widely used in oncology research and is now expanding to other disease states. In addition, a basket design offers benefits over traditional trials, including enabling studies to be conducted over a shorter time period, allowing smaller sample size, and thus, reducing costs.
  In this trial, a parallel Simon two-stage design will be carried out for each basket.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- IBS-D - ORAL-LYO-FMT 7 Weeks (Experimental): Participants with diarrhea-predominant irritable bowel syndrome (IBS-D) receive 7 oral capsules of ORAL-LYO-FMT three times per week (Monday, Wednesday, Friday) for 7 weeks.
  Interventions: Biological: ORAL-LYO-FMT
- IBS-D - Placebo 7 Weeks (Placebo Comparator): Participants with IBS-D receive 7 oral placebo capsules (double-coated and visually identical to active capsules) three times per week for 7 weeks.
  Interventions: Other: Placebo
- IBS-D - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks (Experimental): Participants with IBS-D receive 7 oral capsules of ORAL-LYO-FMT three times per week for 4 weeks, followed by 7 oral placebo capsules three times per week for 3 weeks.
  Interventions: Biological: ORAL-LYO-FMT
- Primary/1st rCDI - ORAL-LYO-FMT 7 Weeks (Experimental): Participants with a primary or first episode of recurrent Clostridioides difficile infection (rCDI) receive 7 oral capsules of ORAL-LYO-FMT three times per week for 7 weeks.
  Interventions: Biological: ORAL-LYO-FMT
- Primary/1st rCDI - Placebo 7 Weeks (Placebo Comparator): Participants with primary or first episode rCDI receive 7 oral placebo capsules three times per week for 7 weeks.
  Interventions: Other: Placebo
- Primary/1st rCDI - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks (Experimental): Participants with primary or first episode rCDI receive 7 oral capsules of ORAL-LYO-FMT three times per week for 4 weeks, followed by placebo capsules three times per week for 3 weeks.
  Interventions: Biological: ORAL-LYO-FMT
- ≥2 rCDI - ORAL-LYO-FMT 7 Weeks (Experimental): Participants with two or more episodes of rCDI receive 7 oral capsules of ORAL-LYO-FMT three times per week for 7 weeks.
  Interventions: Biological: ORAL-LYO-FMT
- ≥2 rCDI - Placebo 7 Weeks (Placebo Comparator): Participants with two or more episodes of rCDI receive 7 oral placebo capsules three times per week for 7 weeks.
  Interventions: Other: Placebo
- ≥2 rCDI - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks (Experimental): Participants with two or more episodes of rCDI receive 7 oral capsules of ORAL-LYO-FMT three times per week for 4 weeks, followed by 3 weeks of placebo capsules.
  Interventions: Biological: ORAL-LYO-FMT

INTERVENTIONS:
Biological: ORAL-LYO-FMT — An oral capsule formulation of lyophilized fecal microbiota. Participants receive 7 capsules, three times per week (Monday, Wednesday, Friday), for either 4 or 7 weeks depending on treatment allocation. The product aims to restore healthy gut microbiota for treatment of IBS-D or prevention of rCDI.
  Arms: IBS-D - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks; IBS-D - ORAL-LYO-FMT 7 Weeks; Primary/1st rCDI - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks; Primary/1st rCDI - ORAL-LYO-FMT 7 Weeks; ≥2 rCDI - ORAL-LYO-FMT 4 Weeks + Placebo 3 Weeks; ≥2 rCDI - ORAL-LYO-FMT 7 Weeks
Other: Placebo — Double-coated oral capsules visually identical to ORAL-LYO-FMT but containing no active material. Participants receive 7 capsules, three times per week, for either 3 or 7 weeks depending on treatment allocation.
  Arms: IBS-D - Placebo 7 Weeks; Primary/1st rCDI - Placebo 7 Weeks; ≥2 rCDI - Placebo 7 Weeks

SUMMARY:
The goal of this clinical trial is to learn if oral lyophilized fecal microbiota therapy (ORAL-LYO-FMT) helps treat diarrhea-predominant irritable bowel syndrome (IBS-D) and prevent the recurrence of Clostridioides difficile infection (rCDI). The main questions it aims to answer are:

* Does ORAL-LYO-FMT reduce IBS symptoms?
* Does it prevent rCDI after treatment?
* What side effects or safety concerns might occur? Researchers will compare ORAL-LYO-FMT to a placebo (a look-alike capsule with no active treatment) to see how well it works.

Participants will:

* Be randomly assigned to take ORAL-LYO-FMT or placebo for up to 7 weeks
* Take capsules three times per week (Monday, Wednesday, Friday)
* Complete health questionnaires and have follow-up visits by phone or in person for up to 6 months The trial also looks at changes in quality of life, mood, and new or ongoing medical conditions over time.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older
* Able to provide informed consent
* Must have at least one of the 3 following conditions:

  1. Irritable bowel syndrome with diarrhea- predominant (IBS-D) as reported by patients of type 6 or 7 in Bristol stool chart and Rome IV diagnostic criteria:

     1. Recurrent abdominal pain/discomfort** at least 3 days/month in last 3 months associated with ≥2 of the following:
     2. Symptom improvement with defecation;
     3. Onset associated with change in stool frequency;
     4. Onset associated with change in stool formation (with this last criterion fulfilled for last 3 months with symptom onset > 6 months prior to diagnosis
  2. Primary or 1 episode recurrent Clostridioides difficile infection which is actively treated with CDI antibiotic (oral vancomycin, oral metronidazole or fidaxomicin) and clinically responding to treatment based on physician assessment at the time of recruitment.
  3. 2 or more episodes of recurrent Clostridioides difficile infection, which is actively treated with CDI antibiotic (oral vancomycin, oral metronidazole or fidaxomicin) and clinically responding to treatment based on physician assessment at the time of recruitment.

Exclusion Criteria:

1. Planned or actively taking other investigational product
2. Unable to tolerate FMT or take oral medications.
3. Requiring systemic antibiotic therapy at the time of FMT
4. Actively taking probiotics [Consumption of yogurt is permitted]
5. Severe allergy to any food and/or medications
6. Major open abdominal surgery within the past 60 days
7. Receipt of chemotherapy or radiation within 8 weeks of screening.
8. Active small bowel obstruction.
9. Those who are pregnant or plan to be pregnant within 3 months of the study. This will be determined on history alone at time of study entry and subsequent follow up.
10. Those who are breastfeeding or plan to breast feed during the trial
11. Not expected to survive beyond 30 days.
12. Any current or previous medical or psychosocial condition or behaviours which in the opinion of the investigator may pose risk to the recipients or the study team

Exclusion Criteria:

-

Ages: 19 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of Recurrent CDI | 8 weeks after completion of IP
  Proportion of participants with Clostridioides difficile infection (CDI) who do not experience recurrence within 8 weeks following completion of the investigational product (IP).
Improvement in IBS Symptom Severity (IBS-SSS) | 8 weeks after completion of IP
  Proportion of IBS-D participants with a reduction in IBS Symptom Severity Score (IBS-SSS) of more than 150 points compared to baseline.

SECONDARY OUTCOMES:
CDI Recurrence Prevention at 24 Weeks | 24 weeks post-treatment
  Proportion of participants with CDI who remain recurrence-free 24 weeks after IP completion.
Longitudinal IBS-SSS Improvement | 1, 3, and 6 months post-treatment
  Proportion of IBS-D participants with sustained improvement in IBS-SSS at 1, 3, and 6 months after IP completion.
Quality of Life (VR-12 Score Change) | Baseline, Week 4, Week 12, and Week 24
  Change in Veterans RAND 12 Item Health Survey (VR-12) scores at baseline, 4 weeks from IP initiation, and 12 and 24 weeks post-IP.
Hospital Anxiety and Depression Scale (HADS) | Baseline, Week 4, Week 12, and Week 24
  Change in HADS scores from baseline to 4, 12, and 24 weeks post-IP.
Chronic Condition Changes | 24 weeks after completion of IP
  Proportion of participants with onset of new or improvement in existing chronic conditions, as reported in long-term follow-up questionnaire.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 8 weeks after completion of IP
  Number and severity of AEs or SAEs possibly or definitely related to IP, assessed via Naranjo Causality Assessment Scale.